CLINICAL TRIAL: NCT00090961
Title: A Randomized Trial Assessing the Effects of Exercise on Patients With Locally Advanced Lung Cancer Undergoing Curative Intent Combined Modality Therapy
Brief Title: S0229, Pulmonary Rehabilitation Education w/wo Exercise Training in Improving Physical Function in Patients Who Are Undergoing Chemo & RT for Locally Advanced Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed early due to poor accrual.
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CDR0000380928; U10CA012027 (NIH); SWOG-S0229
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Lung Cancer; Pulmonary Complications
Keywords: pulmonary complications; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 12-week exercise program + education (Experimental): A 12-week supervised exercise program consisting of 3 days a week on a stationary bike or treadmill. In addition, at the time of enrollment patients are provided educational materials focusing on breathing and energy conservation.
  Interventions: Other: educational intervention; Other: supervised exercise program
- Education (Other): At the time of enrollment patients are provided educational materials focusing on breathing and energy conservation.
  Interventions: Other: educational intervention

INTERVENTIONS:
Other: educational intervention
Other: supervised exercise program
  Arms: 12-week exercise program + education

SUMMARY:
RATIONALE: Pulmonary rehabilitation education and exercise training may improve physical function and quality of life in patients who are receiving treatment for lung cancer.

PURPOSE: This randomized clinical trial is studying pulmonary rehabilitation education and exercise training to see how well they work compared to exercise training alone in improving physical function and quality of life in patients who are undergoing chemotherapy and radiation therapy for locally advanced lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare improvement in physiologic function, in terms of exercise tolerance, in patients with inoperable locally advanced lung cancer undergoing chemoradiotherapy and randomized to pulmonary rehabilitation comprising education with vs without supervised exercise training.
* Compare the health-related quality of life, in terms of multidimensional functioning and patient perception of respiratory difficulties, in patients undergoing these pulmonary rehabilitation interventions.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to Zubrod performance status (0-1 vs 2); FEV_1 (≥ 70% of predicted vs < 70% of predicted); and smoking status* (never smoked or former smoker vs current smoker). Approximately 20 weeks into treatment on SWOG-S0023, patients are randomized to 1 of 2 intervention arms.

NOTE: * Never smoked is defined as < 100 cigarettes in a lifetime and former smoker is defined as no smoking for ≥ 1 year.

* Arm I: Patients participate in a supervised structured exercise program (i.e., walking on a treadmill OR using a stationary exercise bicycle) 3 times a week for 12 weeks. Patients also receive educational materials on how to improve breathing and conserve energy.
* Arm II: Patients receive educational materials as in arm I. In both arms, patients undergo exercise testing using 6-minute walks to measure exercise tolerance at initial evaluation (after randomization but prior to intervention), 12 weeks, and then at 6 and 9 months.

In both arms, intervention continues in the absence of disease progression or the development of other medical conditions that would preclude study participation.

Quality of life is assessed at baseline, 12 weeks, and then at 6 and 9 months.

PROJECTED ACCRUAL: A total of 164 patients (82 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed single, primary bronchogenic lung cancer

  * Inoperable, locally advanced disease (unresectable stage IIIA OR stage IIIB disease)
* The following histologies are eligible:

  * Adenocarcinoma
  * Large cell carcinoma
  * Squamous cell carcinoma
  * Non-lobar and non-diffuse bronchoalveolar carcinoma
  * Small cell lung cancer
* Must have received chemotherapy (platinum based) and radiotherapy for locally advanced unresectable lung cancer

  * Must have achieved a complete response, partial response, or stable disease after treatment

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No acute EKG changes, arrhythmia, or other cardiac abnormality that would preclude study participation
* No uncontrolled cardiac disease
* No recent myocardial infarction

Pulmonary

* Any FEV_1 level by pulmonary function testing

Other

* Willing to participate in 12-week long exercise program
* Chemotherapy-induced neuropathy ≤ grade 2
* No uncontrolled diabetes mellitus
* No other medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2004-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Exercise tolerance | Baseline and at 6 months
  comparison between the control and intervention arms in the percent change in the 6-minute walk distance between baseline and 6 months.

SECONDARY OUTCOMES:
Health-related quality of life | Baseline and at 6 months.
  The difference in total score between pre-study and 6 months for the FACT-L Quality of Life measure.

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette J. Wozniak, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (60):
- United States (60):
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming